CLINICAL TRIAL: NCT00480948
Title: Effects of InFat™ Product (High Sn-2 Palmitic Acid) on Stool Biochemistry and Stool Characteristics in Formula-fed Term Chinese Infants: a Triple-blind, Randomized, Placebo-controlled Trial
Brief Title: Effects of InFat™ Product on Stool Biochemistry and Stool Characteristics in Formula-fed Term Chinese Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study design changes were needed due to change of protocol to a multisite trial and updated set up
Sponsor: Enzymotec (Industry)
Responsible Party: Yael Lifshitz PhD, Enzymotec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: InFat™001
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: infant; infant formula; fatty acids; palmitic acid; stool; calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Infant formula with InFat™ oil(containing ~49% of C16:0 at sn-2 position).
  Interventions: Behavioral: Infant formula feeding (InFat™)
- 2 (Placebo Comparator): Standard vegetable oil based infant formula
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Behavioral: Infant formula feeding (InFat™) — Infant formula with InFat™ oil (containing ~49% of C16:0 at sn-2 position), 24 wk
  Arms: 1
Dietary Supplement: Control — Standard vegetable oil based infant formula
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of infant formula having proportion of palmitate in the sn-2 position comparable to human milk in Chinese term infants.

DETAILED DESCRIPTION:
In human breast milk, and in most infant formulas more than 98% of this milk fat is in the form of triglycerides, which contain saturated and unsaturated fatty acids esterified to glycerol. Fatty acids in human milk-fat have a highly specific positional distribution on the glycerol backbone and this specific configuration is known to have a major contribution to the efficacy of this nutrient absorption.

Palmitic acid (C16:0), the major saturated fatty acid, is predominantly esterified to the sn-2 (β) position of the triglyceride in human milk. In contrast, palmitic acid in standard infant formulas is esterified to the sn-1 and sn-3 positions.

Infants fed with high sn-2 palmitic acid formula had softer stools, less constipation and better calcium absorption as compared to standard infant formula.

InFat™ is structured triglyceride fat ingredient with high levels of palmitic acid at sn-2 position.

The primary objective of this trial is to demonstrate that feeding Chinese term infants, with formula having proportion of palmitate in the sn-2 position comparable to human milk, reduces calcium-soaps formation.

ELIGIBILITY:
Inclusion Criteria:

* Term infants: gestation 37-40 weeks
* Birth weight 2500-4000 g
* Apparent good health
* The infant is a product of normal pregnancy and delivery.

Exclusion Criteria:

* Any maternal disease (psychological or disabled) or socioeconomic problems that may interfere with the mother's ability to take care of her infant
* Major congenital abnormality or chromosomal disorder with a clinical significance that can be detected at birth, clinically significant
* Disease requiring mechanical ventilation or medication treatment at the first week (not including photo treatment for infantile hepatitis)
* Born with a 5- or 10-minute Apgar score <7
* Any suspected or known metabolic or physical limitations interfering with feeding or normal metabolism (require a special formula)
* Breast-feeding for a week or over.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Stool biochemistry - soaped fatty acids | 6 weeks

SECONDARY OUTCOMES:
Stool biochemistry - total fatty acids and calcium content | 6 weeks
Stool characteristics - 7days diaries | 3 months
General health | 3 months
Anthropometric parameters | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi Xiang Su, MD Professor, Principal Investigator — Sun Yat-sen University; Yuming Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat Sen University, Guangzhou, China